CLINICAL TRIAL: NCT06689501
Title: Investigating the Effect of the Combination of L-carnitine Tartrate, Dihydrocapsiate and Protein Yeast Hydrolysate (DNF10) for 12 Weeks on Energy Intake and Energy Expenditure in Overweight and Obese Adults: A Randomised Controlled Trial- (SPICE)
Brief Title: 12-Week Trial Investigating L-carnitine Tartrate, Dihydrocapsiate and Protein Yeast Hydrolysate on Energy Intake and Expenditure in Overweight Adults
Acronym: SPICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Imperial College London (Other); Imperial Clinical Trials Unit (ICTU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2402CLI
Record Dates: First submitted 2024-10-23; First posted 2024-11-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A single-centre, double-blind, placebo-controlled, 2-arm, 12-week trial with randomisation to either the study product (blend of ingredients composed of L-carnitine tartrate, dihydrocapsiate and protein yeast hydrolysate) or placebo.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator)
  Interventions: Combination Product: SPICE BLEND CAPSULE
- Placebo-control arm (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: SPICE BLEND CAPSULE — The study product is a powder mix of L-carnitine tartrate yeast protein hydrolysate and dihydrocapsiate.in the format of hard vegetable green capsules. Participants will consume a total of 4 capsules a day split in two servings.
  Arms: Intervention Arm
Other: Placebo — The matching placebo is microcrystalline cellulose in the format of hard vegetable green capsules. Participants will consume a total of 4 capsules a day split in two servings.
  Arms: Placebo-control arm

SUMMARY:
This is a single-centre, double-blind, randomised, placebo-controlled, 2-arm, parallel-design trial.

This trial will examine the impact of a combined treatment of L-carnitine tartrate, dihydrocapsiate and protein yeast hydrolysate (otherwise known as the "study product") over 12 weeks on energy intake and expenditure in overweight and obese adults.

Approximately 44 participants will be recruited to this trial. Participants will give consent to investigator sites to collect their data. The participants will either be randomised to take the study product or placebo.

The main question that this trial aims to answer is:

The effect of the study product (L-carnitine tartrate, dihydrocapsiate and protein yeast hydrolysate) as compared to placebo on mean energy intake via 3 x 24h dietary recalls online at week 4.

DETAILED DESCRIPTION:
Obesity is a global public health issue that is linked with multiple diseases affecting the body such as the heart, lungs, digestion and metabolism. There are many factors to weight gain that can lead to overweight or obesity. One of them is when more calories (energy for the body from food and drink) are taken in than being used. Weight re-gain of 30-50% of the weight loss occurs within 1 year and 50% of the patients will return to their baseline weight 5 years after they started their weight loss regime. Weight re-gain after weight loss remains an unmet medical need.

This is a single-centre, double-blind, placebo-controlled, 2-arm, 12-week trial with randomisation to either the study product or placebo. The study product is blend of ingredients composed of L-carnitine tartrate, dihydrocapsiate and protein yeast hydrolysate (DNF-10®). Participants will consume a total of 4 capsules a day during 2 different intake occasions. The matching placebo is microcrystalline cellulose.

Ingredients within the study product have individually shown to increase energy expenditure, decrease energy intake, decrease body weight and/or fat mass and decrease appetite in humans, via different pathways. However, they have never been studied in combination. With the combination of these ingredients, Investigator hypothesises the increase of the size effect on negative energy balance via decreasing appetite/energy intake and increasing energy expenditure, targeting different pathways, to >100 kcal/day.

Study participants will provide written informed consent prior to any trial procedures taking place. Participants will attend clinic at the study site 4 times in total as well as complete a validated online questionnaire called Intake24 about foods they've eaten between the in-person study visits.

Main trial procedures include, blood sample collection, online 3x24h dietary recall completion, subjective appetite feelings via 100mm visual analogue scale (VAS) for hunger, fullness, satiety and desire to eat, ad libitum energy intake, energy expenditure (including fat oxidation) using indirect calorimetry, anthropometric measures and administration/compliance to treatment.

ELIGIBILITY:
Inclusion Criteria

1. Aged 21-65 years old (inclusive)
2. Male and Female
3. Body Mass Index (BMI) 28 - <35kg/m2 western criteria for western subjects or 25 - <32kg/m2 for south-Asian ethnicities
4. Comfortable using technology, such as a smartphone or laptop
5. Written informed consent

Exclusion Criteria

1. On unstable medication in the last 6 months, that may impact trial outcomes (e.g., including antibiotics, steroids or medication affecting thyroid hormones, and gut hormones)
2. Weight change of ≥3 kg in the preceding 6 months
3. Eating behaviour disorders such as emotional, restrained or external eating determined via Dutch Eating Behaviour Questionnaire (DEBQ).
4. On a weight loss regime (defined by actively following a diet such as Atkins, weight watchers, meal replacements, low or very low carbohydrate diet, ketogenic diet, intermediate fasting or enrolled into a governmental health program)
5. Significant restrictions on food intake (i.e., regular breakfast skipping, regular cut on carbohydrates, regular intermitted fasting, increased alcohol consumption beyond units defined in exclusion criteria, diet reducing a specific macronutrient, diet significantly reducing calorie intake, excluding a group of food that was not excluded before).
6. Known food intolerances or allergy to any of the interventional supplemental products (L-carnitine, yeast, dihydrocapsiate (synthetic), peppers, cellulose).
7. Taking any drugs in the past 3 months that are GLP-1 receptor analogues, SGLT-2 inhibitors, any weight loss medications and any of the following drugs: cephaloridine, verapamil, valproic acid, and sulfonylureas, usually acting by competitive inhibition of L-carnitine transport by OCTN2 or drugs that affect outcome of interest, including showing a defect on fat absorption (e.g., Orlistat)
8. Known congenital dysfunction of specific organic cation carnitine transporter OCTN2
9. Anaemia
10. Pregnancy or lactation
11. Chronic metabolic disease (except high cholesterol)
12. History of significant organ dysfunction or disease that affect the primary and secondary outcomes of this trial.
13. Life expectancy less than 1 year
14. Known autoimmune disease or genetic disease (including Glucose-6-phosphate deficiency (G6PD) deficiency)
15. Gastrointestinal upset (such as diarrhoea/constipation in the last 2 weeks, abdominal cramping etc.) or disorders such as Chron's disease or inflammatory bowel syndrome or disorder
16. History and ongoing psychiatric illness that affect the primary and secondary outcomes of this trial.
17. Asthma or chronic lung disease requiring long term medications or oxygen.
18. Chronic infective disease, including tuberculosis, hepatitis B and C; and HIV
19. Cancer, coronary heart disease
20. Subjects with history of hypo- and hyperthyroidism
21. Recent blood donation (<8 weeks)
22. Drink >14 units of alcohol per week on a regular basis
23. Consumption of recreational drugs
24. Current smokers (daily)
25. Medical history of difficulties in tolerating/undergoing study procedures planned in the present study, (e.g., like cannulation)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 44 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Change in mean energy intake | week 0 to week 4
  Change in mean energy intake as measured via three consecutive 24-hour dietary recalls conducted online via Intake24, from week 0 to week 4.

SECONDARY OUTCOMES:
1. ENERGY EXPENDITURE | At Week 4 and 12
  a) Postprandial (following a mixed meal tolerance test via standard breakfast) energy expenditure and substrate oxidation (respiratory quotient, fat and carbohydrate oxidation) at 40 - 60min, 100 - 120mins, 160 - 180 min relative to standard breakfast intake (SP will be taken 30 min before breakfast intake) using indirect calorimetry at week 4 and week 12. Indirect calorimetry is a gold-standard, non-invasive technique which is clinically recommended that calculates energy expenditure and substrate oxidation by measuring pulmonary gas exchange (i.e. their production of carbon dioxide and the oxygen inspired). This allows to calculate rates of energy expenditure and substrate oxidation. Endpoint will be incremental Area Under the Curve (iAUC) at 3h.
1. ENERGY EXPENDITURE | At Week 4 and 12
  b) Overnight fasted energy expenditure and substrate oxidation using indirect calorimetry at week 4 and 12 (-20 - 0 min)
2. ENERGY INTAKE AND APPETITE | At Week 12
  a) Energy intake: via 3 x 24h dietary recall (Intake24h).
2. ENERGY INTAKE AND APPETITE | At Week 4 and 12
  b) Ad libitum energy intake: via ad libitum homogeneous meal at 190 min timepoint at week 4 and 12. Food will be weighted before and after to calculate how much food was consumed and converted to kcal.
2. ENERGY INTAKE AND APPETITE | At Week 4 and 12
  c) Subjective appetite feelings: (individual questions and composite appetite score) via 100mm visual analogue scale (VAS) at -50, -40,15, 30, 60, 90, 120, 180 min relative to breakfast intake at week 4 and 12. The outcomes will be composite appetite score of iAUC3h of hunger, satiety, fullness, and desire to eat.
3. ANTHROPOMETRIC MEASURES | At Week 4 and 12
  a) Body weight: At week 4 and 12. Units of measurement: Kg
3. ANTHROPOMETRIC MEASURES | At Week 4 and 12
  b) Waist circumference: Units of measurement: cm
3. ANTHROPOMETRIC MEASURES | At Week 4 and 12
  c) Body Mass Index (BMI): Units of measurement: kg/m^2
3. ANTHROPOMETRIC MEASURES | At Week 4 and 12
  d) Body composition (bioelectrical impedance): Units of measurement: kg
4. SAFETY PROFILES | At Week 4 and 12
  a) Gastrointestinal side effects: For the endpoint, measured using 100mm scale.
4. SAFETY PROFILES | At Week 4 and 12
  b) Nausea: subjective feelings VAS at -50, -40, 15, 30, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC3h. Measured using 100mm scale.
4. SAFETY PROFILES | At Week 4 and 12
  c) Heart rate: At -50, -40, 15, 30, 45, 60, 90,120, 180 min relative to breakfast intake for the endpoint iAUC3h. Units of measurement: bpm
4. SAFETY PROFILES | At Week 4 and 12
  d) C-reactive protein: At -50 min (fasted) relative to breakfast intake for the endpoint. Units of measurement: mg/L
4. SAFETY PROFILES | At Week 4 and 12
  e) Liver function: At -50 min fasted relative to breakfast intake for the endpoint. Units of measurement: g/l
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  c) Fasting: HbA1c. Units of measurement: mmol/mol
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  d) Fasting: liver function: Units of measurement: g/L
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  e) Fasting: C-Reactive Protein: Units of measurement: mg/L
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  f) Fasting: Blood lipid profile. Units of measurement: mmol/L
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  g) Postprandial: gut hormones (GLP-1 at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement for GLP-1: pM
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  h) Postprandial: gut hormones (PYY at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement for PYY: pM
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  i) Postprandial: gut hormones (Ghrelin) at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h at week 4 and 12. Units of measurement of Ghrelin: pg/mL
5. METABOLIC BLOOD PROFILES | At Week 4 and 12
  j) Postprandial: Glucose at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of glucose: mmol/L
5. METABOLIC BLOOD PROFILES | Week 4 and 12
  k) Postprandial: Insulin at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of Insulin: uU/mL or pM

OTHER OUTCOMES:
Exploratory Endpoint: METABOLIC BLOOD PROFILES | Week 4 and 12
  Postprandial: Gut hormones: Glucose-dependent insulinotropic polypeptide [GIP], Cholecystokinin, Oxyntomodulin) at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement: pM
Exploratory Endpoint: METABOLIC BLOOD PROFILES | Week 4 and 12
  Postprandial: Gut hormone- Leptin at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of Leptin: ng/mL.
Exploratory Endpoint: METABOLIC BLOOD PROFILES | Week 4 and 12
  Postprandial: Gut hormone- CCK at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of CCK:
Exploratory Endpoint: METABOLIC BLOOD PROFILES | Week 4 and 12
  Postprandial: Gut hormone- Adiponectin at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of Adiponectin:
Exploratory Endpoint: METABOLIC BLOOD PROFILES | Week 4 and 12
  Postprandial: Gut hormone: Growth differentiation factor 15 [GDF-15] at -50, -40,15, 30, 45, 60, 90, 120, 180 min relative to breakfast intake for the endpoint iAUC1h and iAUC3h. Units of measurement of GDF-15: pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chambers, Principal Investigator — Imperial College London, Department of Metabolism, Digestion and Reproduction
Locations (1):
- Imperial College Healthcare NHS Trust, Hammersmith Hospital, 72 Du Cane Rd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No